CLINICAL TRIAL: NCT06413485
Title: Canadian Beach Cohort Study: Prospective Study to Assess the Burden of Recreational Water Illness
Brief Title: Canadian Beach Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Toronto Metropolitan University (Other)
Collaborators: University of Waterloo (Other); University of Guelph (Other); Health Canada (Other Government); Public Health Agency of Canada (PHAC) (Other Government); Toronto Public Health (Other Government); Vancouver Coastal Health (Other Government); Government of Manitoba (Unknown); Niagara Region Public Health (Other); McMaster University (Other); Halifax Regional Municipality (Unknown)
Responsible Party: Principal Investigator, Ian Young, Associate Professor, Toronto Metropolitan University
Other Study IDs: PJT-192023
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Water-Related Diseases; Gastrointestinal Diseases
Keywords: Epidemiology; Beach water; Water quality; Fecal pollution; Cohort study; Mixed methods; Environmental health
MeSH Terms: conditions — Waterborne Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Beachgoers: Beachgoing families and households to one or more Canadian beaches during the summers of 2023 to 2026.
  Interventions: Behavioral: Level of recreational water contact activities

INTERVENTIONS:
Behavioral: Level of recreational water contact activities — We will examine a graded classification of this exposure based on individuals' minimum level of water contact: 1) no water contact; 2) minimal contact; 3) body immersion; 4) swallowed water. Minimal contact is defined as water contact that does not result in body immersion (e.g., wading below one's waist, boating, fishing). Body immersion is defined as entering the water above one's waist (e.g., swimming, surfing, snorkelling), and swallowing water as ingestion of any amount of water.
  Other Names: Sand contact at beaches

SUMMARY:
Swimming and other water activities at public beaches are increasingly popular leisure activities among Canadians. However, these activities can lead to increased risks of acquiring acute gastrointestinal illness and respiratory, skin, ear, and eye infections among beachgoers. These illnesses have a significant health and economic burden on society, with young children having much higher rates of illness than other age groups. Currently, baseline data are lacking on the risk of recreational water illness in Canada, and beachgoers may lack awareness and understanding of these risks and how to prevent them. This study will identify the burden of recreational water illness among Canadian beachgoers. The results will be used to develop recommendations for improving recreational water quality guidelines for safe swimming in Canada, as well as public health risk management and communication strategies with beachgoers. The study will use a mixed-methods approach, consisting of a prospective cohort study and a qualitative study of beachgoers. The investigators will determine the risk of acquiring recreational water illness outcomes in beachgoers that engage in different levels of water and sand contact. The investigators will examine differences in illness risks by beachgoer gender, age, and location. The investigators will examine relationships between fecal indicator bacteria (E. coli), environmental conditions, and host-specific biomarkers with the risk of gastrointestinal illness among beachgoers. The investigators will also evaluate beachgoer risk perceptions and behaviours toward recreational water quality. The study will take place at five targeted beach sites in British Columbia, Manitoba, and Ontario. The study will be coordinated by a multidisciplinary research team, with activities guided by a stakeholder steering group consisting of key knowledge users. The long-term goal is to reduce the burden of recreational water illness in Canada, contributing to improved public health.

DETAILED DESCRIPTION:
Swimming and other beach water activities are increasingly popular outdoor leisure activities among Canadians. However, these activities increase the risk of acquiring acute gastrointestinal illness (AGI) and other acute illnesses among beachgoers. Recreational water illness (RWI) has a significant health burden, with young children having the highest rates of illness. These illnesses result in substantial costs to society due to healthcare costs and lost productivity. Data are lacking in Canada on the risk and burden of RWI, and beachgoers may lack awareness and understanding of RWI risks and how to prevent them. There is a critical need to conduct timely research on the burden of RWI in Canada to inform recreational water quality guidelines and public health risk management.

The purpose of this study is to identify the burden of RWI among Canadian beachgoers and to develop recommendations for improving recreational water quality risk management, communication, and pollution source prevention. The objectives are to:

1. Measure the risk and burden of five different RWI outcomes (AGI, respiratory, eye, ear, and skin infections) in beachgoers that engage in different levels of water and sand contact;
2. Identify differences in RWI risks by beachgoer gender, age, and beach location;
3. Determine relationships between fecal indicator bacteria, environmental parameters, host-specific biomarkers, and the risk of AGI among beachgoers; and
4. Understand beachgoer risk perceptions and behaviours related to recreational water quality and socio-political issues that may impact RWI risks among beachgoers.

The study will use a mixed-methods approach, consisting of a prospective cohort study (Objectives 1-3) with embedded qualitative research (Objective 4). The cohort study will involve enrolling participants at public beaches, ascertaining their water and sand contact exposure status, then following-up to determine the incidence of acute RWI outcomes. The investigators will combine beachgoer exposure data with routinely collected secondary data on environmental parameters and E. coli levels in beach water. The investigators will also test for enterococci as another fecal indicator using rapid molecular methods and will conduct microbial source tracking to determine the contribution of different sources of fecal contamination (e.g., human, avian) to AGI. The study will take place at eight targeted freshwater and marine beach sites in British Columbia, Manitoba, and Ontario. The qualitative research will consist of focus groups to determine beachgoer risk perceptions and behaviours toward recreational water quality and key informant interviews with stakeholders to provide additional socio-political insights and context.

The long-term goal of this study is to reduce the burden of RWI in Canada, contributing to improved public health. The study will be led by an experienced, diverse, and multi-disciplinary research team, including engagement with public health and environmental authorities. Activities will be guided by a stakeholder steering group consisting of key knowledge-users (KUs). This integrated KT approach will help to ensure that the results are relevant and useful to KUs, facilitating their direct uptake to influence recreational water quality policies and practice.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent for the study and complete the surveys in English or French
* Home address in Canada or the U.S.
* Must not have participated in the study in the past 21 days

Exclusion Criteria:

* Not a Canadian or U.S. resident.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Beachgoing households and individuals present at one of the targeted study beach sites during the recruitment period.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Acutre gastrointestinal illness (AGI) | Within 7 days of beach visit/water contact
  Self-reported AGI in the 7-day period following beach water contact. Defined as one or more of: (a) diarrhea (≥3 loose stools in 24 hrs); (b) vomiting; (c) nausea with stomach cramps; or (d) nausea or stomach cramps that interfere with regular daily activities (e.g., missed work or school).

SECONDARY OUTCOMES:
Acute respiratory illness | Within 7 days of beach visit/water contact
  Self-reported fever with sore throat, fever with nasal congestion, or cough with phlegm
Skin infection | Within 7 days of beach visit/water contact
  Self-reported rash or itchy skin
Ear infection or earache | Within 7 days of beach visit/water contact
  Self-reported ear infection or earache
Eye infection or irritation | Within 7 days of beach visit/water contact
  Self-reported eye infection or irritation

CONTACTS AND LOCATIONS:
Overall Officials: Ian Young, Principal Investigator — School of Occupational and Public Health, Toronto Metropolitan University
Locations (5):
- Canada (5):
  - English Bay Beach and Kitsilano Beach, Vancouver, British Columbia
  - Grand Beach, Winnipeg, Manitoba
  - Birch Cove Beach, Halifax, Nova Scotia
  - Bay Beach and Nickel Beach, Fort Erie, Ontario
  - Sunnyside and Marie Curtis Park East beaches, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made publicly available following the study conclusion and publication of results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Study protocol will be submitted for publication in 2024, and will contain the analysis plan. The final consent form and code will be shared with publication of the results later in the study timeframe (2027-2028).
URL: https://www.canadianbeachwater.ca/